CLINICAL TRIAL: NCT01591759
Title: A Pilot Trial of Citicoline in Individuals With mTBI
Brief Title: A Pilot Trial of Citicoline in Individuals With Mild Traumatic Brain Injury (mTBI)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Our citicoline supply expired and the exact product has discontinued.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Staci Gruber, Ph.D., Director, Cognitive and Clinical Neuroimaging Core/Assistant Professor of Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCL 2011-P-002028
Record Dates: First submitted 2012-02-29; First posted 2012-05-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Traumatic Brain Injury
Keywords: citicoline; cognitive function; function magnetic resonance imaging; magnetic resonance spectroscopy; diffusion tensor imaging
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citicoline (Experimental): 8-week treatment of 2,000mg/day of citicoline
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citicoline — 2,000mg/day of citicoline taken as twice daily unit doses of 1,000 mg for the 8-week period of the clinical trial
  Other Names: Citicoline Sodium
  Arms: Citicoline
Drug: Placebo — Placebo arm of single-blind study
  Arms: Placebo

SUMMARY:
This investigation will explore the impact of 8 weeks of citicoline treatment on cognitive function, clinical state and substance use in 40 individuals with mild traumatic brain injury (mTBI).

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains a major cause of death and disability within the United States. Approximately 1.4 million individuals sustain a TBI each year, and currently, more than 5.3 million Americans or 3% of the general population live with disabilities associated with a TBI, resulting in enormous financial, physical and psychosocial burdens to the patients, their families and society. The issue of TBI has never been more salient, as it is now labeled the "signature wound" of the current conflict in Iraq and Afghanistan.

Patients with mTBI often experience a variety of symptoms including headache, dizziness, fatigue, irritability, depression, anxiety, insomnia, reduced alcohol tolerance, and problems with cognitive function. In acute stages, cognitive deficits may affect multiple domains and be severe enough to interfere with everyday activities.

The proposed investigation will explore the impact of 8 weeks of citicoline treatment on cognitive function, clinical state and substance use in 40 individuals with mTBI. The investigators hypothesize that individuals with mTBI who receive citicoline will demonstrate improvements in cognitive performance relative to their own pre-treatment levels as well as to those randomized to placebo. Specifically, the investigators expect the greatest improvement on frontal/executive measures following treatment with citicoline. In addition, the investigators also hypothesize that 8 weeks of treatment with citicoline will result in a reduction of comorbid substance use and improvements in clinical state measures relative to both pre-treatment levels and those randomized to receive placebo. Given the relationship between cognitive function and clinical state, the investigators expect a primary improvement in cognitive function will likely precede the expected improvement of mTBI-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent
* Subject is cooperative
* Subject is between 18 and 35 years of age (inclusive)
* Subject meets criteria for mTBI
* Subject has separate treating physician and is willing to provide consent for treating physician to be contacted by research team
* Subject is a native English speaker or acquired English prior to age 5

Exclusion Criteria:

* Serious medical illness, including diabetes, neurodegenerative disorder (i.e. multiple sclerosis, lupus, etc)
* Neurological disorder or history of serious head trauma resulting in loss of extended loss of consciousness or coma
* History of ECT treatment
* Estimated IQ < 75
* Positive urine pregnancy test (screened on all study visits)

Additional MR Imaging Exclusion Criteria:

* Presence of a medical condition known to affect MR BOLD imaging (i.e. metabolism disorders, eating disorders, hormonal dysregulation, etc)
* Uncorrectable poor vision, as subjects must have normal or corrected-to normal vision for viewing of cognitive challenge paradigms during fMRI protocols
* Claustrophobia or metal implanted within the body, including body piercings which are not removable
* Additional MR related contraindications:

  * Cardiac pacemakers
  * Metal clips on blood vessels (also called stents)
  * Artificial heart valve, artificial arms, hands, legs, etc.
  * Brain stimulator devices
  * Implanted drug pumps
  * Ear or eye implants
  * Known metal fragments in eyes
  * Exposure to metal filings (sheetmetal workers, welders, and others)
  * Other metallic surgical hardware in vital area
  * Certain tattoos with metallic ink
  * Certain transdermal (skin) patches such as:
  * NicoDerm (nicotine for tobacco dependence)
  * Transderm Scop (scopolamine for motion sickness)
  * Ortho Evra (birth control)
  * Certain intrauterine devices (IUDs containing metal)
* Since some will be military veterans with combat experience and may have been exposed to shrapnel, they will be screened with a handheld metal detector to ensure that they do not have any metal embedded in their body. Subjects who do not pass the metal detector screen and subjects with known shrapnel or other metal embedded or implanted in their body will not be eligible to participate in the MRI portion of this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Assessment Changes with Citicoline Treatment | At baseline and at treatment week 4 and week 8
  4-Subtest Wechsler Abbreviated Scale of Intelligence (WASI) at the baseline visit only. Measures to be administered at baseline and both follow-up visits: Hopkins Verbal Learning Test-Revised (HVLT-R), Brief Visuospatial Memory Test-Revised (BVMT-R), Logical Memory (LM) Subtest of the Wechsler Memory Scale-Revised (WMS-R) and Sullivan Multiple Versions, Rey-Osterreith Complex Figure (Rey-O), Stroop Color-Word Test, Trailmaking Test A & B, Controlled Oral Word Association Test (COWAT), Digit Span subtest of the WAIS-R, Digit Symbol Substitution Test (DSST), Wisconsin Card Sort Test (WCST), Go/No Go Test, Time Estimation Task (TET), and Facial Expressions of Emotion-Stimuli and Tests (FEEST).

SECONDARY OUTCOMES:
Clinical State Assessment Changes with Citicoline Treatment | Weekly assessment & biweekly clinical scales for 8 weeks
  Montgomery-Asberg Depression Rating Scale (MADRS), Young Mania Rating Scale (YMRS), Hamilton Anxiety Scales (HAM-A), Positive & Negative Affect Scale (PANAS), Profile of Mood States (POMS), Barratt Impulsiveness Scale (BIS), UPPS Impulsive Behavior Scale (UPPS-P), Impulsiveness-Venturesomeness-Empathy Scale (IVE), State/Trait Inventory (STAI), Beck Depression Inventory (BDI), Beck Hopelessness Scale (BHS), Beck Scale for Suicidal Ideation (BSS), Beck Anxiety Inventory (BAI), Frontal Systems Behavior Scale (FrSBe), Alcohol Use Disorders Identification Test (AUDIT), Cannabis Use Disorders Identification Test-Revised (CUDIT-R), National Center for PTSD 17-item checklist (PCL), Neurobehavioral Symptom Inventory (NSI), Combat Exposure Scale (CES), & Clinician Administered PTSD Scale (CAPS).
Functional MRI and Diffusion Tensor Imaging Changes with Citicoline Treatment | At baseline and at treatment week 8
  All functional MR imaging (fMRI) will be performed on the 3 Tesla (3T) scanner retrofitted with a whole body echo-planar coil with a TIM upgrade. The challenge paradigms will be a Masked Affect paradigm, the Multi-Source Interference Task (MSIT), and a Trauma-Related Emotional Counting Stroop. In addition, diffusion tensor imaging (DTI) will be acquired to assess white matter microstructure integrity by measuring fractional anisotropy (FA) and mean diffusivity (MD).
Magnetic Resonance Spectroscopy Changes with Citicoline Treatment | At baseline and at treatment week 8
  Proton magnetic resonance spectroscopy (MRS) will be acquired at 3 Tesla using both single voxel and chemical shift imaging (CSI) techniques in order to assess brain metabolite levels pre and post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Staci A Gruber, Ph.D., Principal Investigator — Mclean Hospital; Scott E Lukas, Ph.D., Study Chair — Mclean Hospital
Locations (1):
- McLean Hospital Brain Imaging Center, Belmont, Massachusetts, United States